CLINICAL TRIAL: NCT01379963
Title: Non-interventional Study of Six-month Retrospective Reporting of Hemoglobin Levels in Patients With Renal Anaemia Who Are Treated With MIRCERA® (Methoxy-polyethylene-glycol-epoetin Beta)
Brief Title: A Retrospective Observational Study of Hemoglobin Levels in Patients With Renal Anemia Treated With Mircera (Methoxy Polyethylene Glycol-Epoetin Beta)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22014
Record Dates: First submitted 2011-06-22; First posted 2011-06-23 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-05

CONDITIONS: Anemia, Kidney Disease, Chronic
MeSH Terms: conditions — Anemia; Kidney Diseases; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This retrospective observational study will evaluate the hemoglobin levels in patients with renal anemia over 6 months treatment with Mircera (methoxy polyethylene glycol-epoetin beta).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Renal anemia treated with Mircera for at least 6 months before entering study

Exclusion Criteria:

* Patients who refuse or are incapable of giving their written informed consent to retrospective data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with renal anemia on treatment with Mircera
Sampling Method: Probability Sample
Enrollment: 780 (Actual)
Dates: Start 2009-04-30 (Actual); Primary Completion 2011-02-28 (Actual); Study Completion 2011-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Greece (17):
  - Timios Stavros Clinic; Nephrology Department, Aigáleo
  - General Hospital of Artas; Nephrology, Arta
  - Pantokrator Private Clinic; Nephrology, Athens
  - Attikon Center; Nephrology, Athens
  - Athinaiki Private Clinic, Athens
  - Kyanos Stavros Private Hospital; Nephrologic Clinic, Athens
  - Iaso General Private Clinic; Nephrology, Athens
  - Iatriko Athinon Clinic Dafnis; Nephrology Department, Daphni-athens
  - Kyanous Stavros of Patras, Renal Disease Therapy Unit, Pátrai
  - Olympion Therapeytirion; Nefrology, Pátrai
  - Iasis Private Clinic, Piraeus
  - General Hospital Of Chalkidikis; Dialysis Center Unit, Polygyros
  - Diavalkaniko Kentro; Nephrology, Thessaloniki
  - General Hospital of Thessalonikis G.Papanikolaou; Nephrology, Thessaloniki
  - Alfa Nefrodynamiki; Nefrology, Thessaloniki
  - Thessaliki Nossileytiki; Nephrology, Volos
  - General Hospital of Volos; Nephrology, Volos

RESULTS

PARTICIPANT FLOW:
Groups:
- Methoxy-Polyethylene-Glycol-Epoetin Beta: Participants with renal anemia who were treated with methoxy-polyethylene-glycol-epoetin beta (Mircera, Continuous Erythropoietin Receptor Activator [C.E.R.A]) according to the standard clinical practice, were observed for at least 6 months in this retrospective study.
Period: Overall Study
Arm/Group | Methoxy-Polyethylene-Glycol-Epoetin Beta
Started | 780
Completed | 780
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all enrolled participants.
Groups:
- Methoxy-Polyethylene-Glycol-Epoetin Beta: Participants with renal anemia who were treated with methoxy-polyethylene-glycol-epoetin beta according to the standard clinical practice, were observed for at least 6 months in this retrospective study.
Arm/Group | Methoxy-Polyethylene-Glycol-Epoetin Beta
Number analyzed (Participants) | 780
Age, Continuous [Mean (Standard Deviation); unit: Years] — Here, 773 participants were analyzed for this baseline measure (age). Since this is a non-interventional retrospective study participants with missing data were excluded from the analysis.
  Years | 68.64 (14.10)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 442
  Male | 325
  Missing | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a 3-month Hemoglobin Level Stabilization in the Range of 11-12 Grams Per Deciliter (g/dL)
Description: Hemoglobin level stabilization within the range of 11-12 g/dL was measured on a monthly basis according to Kidney Disease Outcomes Quality Initiative (KDOQI) guidelines, for enrolled participants who had received methoxy-polyethylene-glycol-epoetin beta treatment.
Time Frame: Up to 6 months
Population: Analysis population included all enrolled participants who had received study treatment and were monitored for hemoglobin level on a monthly basis, according to standard clinical practice. Here, number of participants analyzed signifies those participants who were evaluable for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy-Polyethylene-Glycol-Epoetin Beta
Number analyzed (Participants) | 774
Percentage of participants | 17.18

2. Secondary Outcome: Percentage of Participants Who Achieved a 6-month Hemoglobin Level Stabilization in the Range of 11-12 g/dL
Description: Hemoglobin level Level stabilization within the range of 11-12 g/dL was measured on a monthly basis according to KDOQI guidelines, for enrolled participants who had received methoxy-polyethylene-glycol-epoetin beta treatment.
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy-Polyethylene-Glycol-Epoetin Beta
Number analyzed (Participants) | 776
Percentage of participants | 3.09

ADVERSE EVENTS:
Description: This was a retrospective study, so the adverse events have already been reported according to the current pharmacovigilance regulations. In addition, this study did not aim to evaluate the safety of methoxy-polyethylene glycol-epoetin beta.
Arm/Group | Methoxy-Polyethylene-Glycol-Epoetin Beta
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigators is free to publish in reputed journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.